CLINICAL TRIAL: NCT03649360
Title: Knee Pain After Tibial Shaft Fracture Treated With Intramedullary Nailing
Brief Title: Knee Pain After Intramedullary Nailing in the Tibia
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Nikolaj Erin-Madsen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: IMN Study
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Tibia Fracture; Knee Pain Chronic
Keywords: Knee pain; Intramedullary tibial nail; KOOS
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to evaluate the long-term outcome after inserting an intramedullary nail in patients with a tibial shaft fracture using an injury-specific questionnaire.

DETAILED DESCRIPTION:
Introduction

The treatment of choice for unstable diaphyseal fractures in the tibia is reamed insertion of an intramedullary nail (IMN) with the additional placement of interlocking screws. The most common complication after insertion of an IMN as treatment of tibial shaft fractures is chronic knee pain with reported rates between 10 % and 87 % with a mean of 47,4 % in metaanalyses.

Methods

The primary objective of this study is to evaluate the long-term outcome after inserting an IMN in patients with a tibial shaft fracture using an injury-specific questionnaire.

This study includes patients operated on five Danish hospitals. A database search was made using operational codes for insertion of an IMN in a five-year period. Patients aged 18 years or older, alive and residing in Denmark at the time of follow-up could be included in the study. These patients then received a Knee Injury and Osteoarthritis Score (KOOS) questionnaire by mail with questions regarding knee-specific symptoms, stiffness, pain, function and quality of life. Questionnaires were filled out and returned to the corresponding physician for further analyze. Patients who were unable to fill out the questionnaire due to concomitant physical condition or who had undergone amputation or further surgery on the affected limb were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, alive and residing in Denmark at the time of follow-up could be included in the study.

Exclusion Criteria:

* Patients who were unable to fill out the questionnaire due to concomitant physical condition or who had undergone amputation or further surgery on the affected limb were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent surgery with reamed, locked intramedullary nailing after isolated tibial shaft fracture at one of the above mentioned orthopedic departments between 1st of November 2009 and 30th of October 2014 were sought.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Knee Pain after Tibial Shaft Fracture Treated with Intramedullary Nailing | 1st of November 2009 till 30th of October 2014.
  The primary objective of this study is to evaluate the long-term outcome after inserting an IMN in patients with a tibial shaft fracture using an injury-specific questionnaire. We used the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire to collect patient data. It is used to assess patient's subjective opinion about symptoms related to the knee and other associated problems. The questionnaire has been translated and validated in Danish and consists of 5 subscales: pain, symptoms, function in daily living (ADL) function in sports and recreation and knee-related QOL. Each subscale has between 4 and 17 questions (a total of 42 questions) with each question having 5 options ranging from no symptoms to severe symptoms. Each question gets a score from 0-4 and a score from 0-100 is calculated. 100 indicating no symptoms and 0 indicates major symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Erin-Madsen, MD, Study Director — Copenhagen University Hospital of Hvidovre
Locations (1):
- Copenhagen University Hospital of Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan of sharing data.

REFERENCES:
- [Background] Bone LB, Johnson KD. Treatment of tibial fractures by reaming and intramedullary nailing. J Bone Joint Surg Am. 1986 Jul;68(6):877-87. PMID 3733776
- [Background] Bone LB, Sucato D, Stegemann PM, Rohrbacher BJ. Displaced isolated fractures of the tibial shaft treated with either a cast or intramedullary nailing. An outcome analysis of matched pairs of patients. J Bone Joint Surg Am. 1997 Sep;79(9):1336-41. doi: 10.2106/00004623-199709000-00007. PMID 9314395
- [Background] Court-Brown CM, Gustilo T, Shaw AD. Knee pain after intramedullary tibial nailing: its incidence, etiology, and outcome. J Orthop Trauma. 1997 Feb-Mar;11(2):103-5. doi: 10.1097/00005131-199702000-00006. PMID 9057144
- [Background] Hiesterman TG, Shafiq BX, Cole PA. Intramedullary nailing of extra-articular proximal tibia fractures. J Am Acad Orthop Surg. 2011 Nov;19(11):690-700. doi: 10.5435/00124635-201111000-00005. PMID 22052645
- [Background] Lefaivre KA, Guy P, Chan H, Blachut PA. Long-term follow-up of tibial shaft fractures treated with intramedullary nailing. J Orthop Trauma. 2008 Sep;22(8):525-9. doi: 10.1097/BOT.0b013e318180e646. PMID 18758282
- [Background] Toivanen JA, Vaisto O, Kannus P, Latvala K, Honkonen SE, Jarvinen MJ. Anterior knee pain after intramedullary nailing of fractures of the tibial shaft. A prospective, randomized study comparing two different nail-insertion techniques. J Bone Joint Surg Am. 2002 Apr;84(4):580-5. doi: 10.2106/00004623-200204000-00011. PMID 11940618
- [Background] Karladani AH, Granhed H, Edshage B, Jerre R, Styf J. Displaced tibial shaft fractures: a prospective randomized study of closed intramedullary nailing versus cast treatment in 53 patients. Acta Orthop Scand. 2000 Apr;71(2):160-7. doi: 10.1080/000164700317413139. PMID 10852322
- [Background] Morandi M, Banka T, Gaiarsa GP, Guthrie ST, Khalil J, Hoegler J, Lindeque BG. Intramedullary nailing of tibial fractures: review of surgical techniques and description of a percutaneous lateral suprapatellar approach. Orthopedics. 2010 Mar;33(3):172-9. doi: 10.3928/01477447-20100129-22. No abstract available. PMID 20205366
- [Background] Karachalios T, Babis G, Tsarouchas J, Sapkas G, Pantazopoulos T. The clinical performance of a small diameter tibial nailing system with a mechanical distal aiming device. Injury. 2000 Jul;31(6):451-9. doi: 10.1016/s0020-1383(00)00024-3. PMID 10831746
- [Background] Katsoulis E, Court-Brown C, Giannoudis PV. Incidence and aetiology of anterior knee pain after intramedullary nailing of the femur and tibia. J Bone Joint Surg Br. 2006 May;88(5):576-80. doi: 10.1302/0301-620X.88B5.16875. No abstract available. PMID 16645100
- [Background] Vaisto O, Toivanen J, Kannus P, Jarvinen M. Anterior knee pain after intramedullary nailing of fractures of the tibial shaft: an eight-year follow-up of a prospective, randomized study comparing two different nail-insertion techniques. J Trauma. 2008 Jun;64(6):1511-6. doi: 10.1097/TA.0b013e318031cd27. PMID 18545115
- [Background] Althausen PL, Neiman R, Finkemeier CG, Olson SA. Incision placement for intramedullary tibial nailing: an anatomic study. J Orthop Trauma. 2002 Nov-Dec;16(10):687-90. doi: 10.1097/00005131-200211000-00001. PMID 12439190
- [Background] Weninger P, Schultz A, Traxler H, Firbas W, Hertz H. Anatomical assessment of the Hoffa fat pad during insertion of a tibial intramedullary nail--comparison of three surgical approaches. J Trauma. 2009 Apr;66(4):1140-5. doi: 10.1097/TA.0b013e318169cd4d. PMID 19359927
- [Background] Hernigou P, Cohen D. Proximal entry for intramedullary nailing of the tibia. The risk of unrecognised articular damage. J Bone Joint Surg Br. 2000 Jan;82(1):33-41. doi: 10.1302/0301-620x.82b1.9818. PMID 10697311
- [Background] Orfaly R, Keating JE, O'Brien PJ. Knee pain after tibial nailing: does the entry point matter? J Bone Joint Surg Br. 1995 Nov;77(6):976-7. No abstract available. PMID 7593119
- [Background] Bhattacharyya T, Seng K, Nassif NA, Freedman I. Knee pain after tibial nailing: the role of nail prominence. Clin Orthop Relat Res. 2006 Aug;449:303-7. doi: 10.1097/01.blo.0000223976.91089.08. PMID 16702914
- [Background] Ryan SP, Tornetta P 3rd, Dielwart C, Kaye-Krall E. Knee pain correlates with union after tibial nailing. J Orthop Trauma. 2011 Dec;25(12):731-5. doi: 10.1097/BOT.0b013e318213f587. PMID 21886000
- [Background] Demirtas A, Azboy I, Durakbasa MO, Ucar BY, Mercan AS, Cakir IA. [The relationship between the quadriceps muscle strength and the anterior knee pain occurring after locked intramedullary nailing for tibial diaphysis fractures]. Eklem Hastalik Cerrahisi. 2011 Aug;22(2):81-4. Turkish. PMID 21762062
- [Background] Vaisto O, Toivanen J, Kannus P, Jarvinen M. Anterior knee pain and thigh muscle strength after intramedullary nailing of a tibial shaft fracture: an 8-year follow-up of 28 consecutive cases. J Orthop Trauma. 2007 Mar;21(3):165-71. doi: 10.1097/BOT.0b013e31803773cd. PMID 17473752
- [Background] Weller S, Kuner E, Schweikert CH. Medullary nailing according to Swiss study group principles. Clin Orthop Relat Res. 1979 Jan-Feb;(138):45-55. PMID 445918
- [Background] Lottes JO. Medullary nailing of the tibia with the triflange nail. Clin Orthop Relat Res. 1974 Nov-Dec;(105):53-66. No abstract available. PMID 4609657
- [Background] Paradowski PT, Bergman S, Sunden-Lundius A, Lohmander LS, Roos EM. Knee complaints vary with age and gender in the adult population. Population-based reference data for the Knee injury and Osteoarthritis Outcome Score (KOOS). BMC Musculoskelet Disord. 2006 May 2;7:38. doi: 10.1186/1471-2474-7-38. PMID 16670005
- [Derived] Erin-Madsen N, Aasvang TK, Viberg B, Bloch T, Brix M, Tengberg PT. Knee pain and associated complications after intramedullary nailing of tibial shaft fracture. Dan Med J. 2019 Aug;66(8):A5554. PMID 31315794
- See also: KOOS questionnaire [KOOS web site]. Accessed May 20th 2015. — http://www.koos.nu
- See also: Danish Database of Fractures website. Accessed March 25, 2015. — http://www.DFDB.dk